CLINICAL TRIAL: NCT02054975
Title: Prospective Open Pilot of Low vs. Higher Dose Vitamin D in D-deficient Asthmatic Children: Does Diet Predict Immune Function and Asthma Symptom Response to Vitamin D Supplementation?
Brief Title: Vitamin D in Pediatric Asthma: a Randomized Controlled Open-label Pilot Trial
Acronym: D-Asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nationwide Children's Hospital (Other)
Collaborators: Ohio State University (Other)
Responsible Party: Principal Investigator, Barbara Gracious, Principal Investigator, Nationwide Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB13-00504
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Asthma; Vitamin D Deficiency
Keywords: asthma, children, vitamin D deficiency, clinical trial
MeSH Terms: conditions — Asthma; Vitamin D Deficiency | interventions — Ergocalciferols; Cholecalciferol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- vitamin D2 + vitamin D3 (Experimental): Vitamin D2 50,000 IU each week x 4 + vitamin D3 4,000 IU each day for 3 months
  Interventions: Drug: Vitamin D2 + vitamin D3
- Vitamin D lower dose (Active Comparator): 800 IU vitamin D3 by mouth each day for 3 months
  Interventions: Drug: Vitamin D3

INTERVENTIONS:
Drug: Vitamin D2 + vitamin D3 — higher dose vitamin D
  Other Names: Vitamin D2 50,000 IU by mouth once per week x 4 weeks; Vitamin D3 4,000 IU by mouth once each day
  Arms: vitamin D2 + vitamin D3
Drug: Vitamin D3 — lower dose vitamin D
  Other Names: Vitamin D3 800 IU by mouth each day for 3 months
  Arms: Vitamin D lower dose

SUMMARY:
This is a pilot randomized controlled trial of lower vs. higher dose vitamin D supplementation in D-deficient asthmatic children, to determine necessary sample sizes for outcome measures in a larger multisite study, and to examine possible relationships and effect sizes between various biological markers that may be important to the pathophysiology of childhood asthma.

Aims of the study are to:

1. Evaluate effect sizes for relationships between serum 25OH-vitD and omega-fatty acid (FA) biomarkers, before and after supplementation with lower or higher dose vitamin D, on immune function, and asthma severity.
2. Characterize changes in innate and adaptive immune function and inflammatory responses in asthmatic D-deficient youth at baseline and after vitD supplements, by dietary O6:O3FA status and vitD dose.

DETAILED DESCRIPTION:
An estimated up to 120 youth meeting eligibility criteria will be screened for vitamin D deficiency, and if found deficient, will be offered enrollment in this study.

Eligible children who assent and whose parent/guardian consent to participate will be randomized to low dose vs. higher dose vitamin D to take across a 3-month period of time. Blood, questionnaires, and pulmonary function tests will be obtained at baseline and end of study. Weekly phone calls will check on any questions or concerns the participant or their family may have.

Aims and Hypotheses:

Aim I: Evaluate effect sizes for relationships between omega-FA and vitD biomarkers, pre- and post- low and higher dose vitamin D supplementation, in diet, immune function, and asthma severity.

Aim II: Characterize changes in innate and adaptive immune function and inflammatory responses in asthmatic D-deficient youth at baseline and after vitD supplements, by O6:O3FA status and vitD dose.

Exploratory: Compute effect sizes/odds ratios for differences in pulmonary function, self-reported asthma severity, depressive symptoms, hospitalization/ED visits, and medication changes based on treatment group.

Effect sizes will be calculated for all continuous outcome variables by:

Effect Size (ES) = Average of the post-test scores - Average of the pre-test scores Average standard deviation

Odds ratios for the categorical asthma severity variable will be computed through logistic regression by treatment group with no covariates.

Examine differences in pulmonary function tests, self-reported asthma severity, depressive symptoms, hospitalization/ED visits, and medication changes based on treatment group. Omega fatty acid intake and allergic status will be included as potentially mediating variables.

ELIGIBILITY:
Inclusion Criteria:

* 1. Informed consent and assent signed and dated before participation.
* 2. Male or female, ages 8 through 17 at baseline; all races and ethnicities
* 3. asthma and currently taking a prescribed daily inhaled steroid asthma medication
* 4. English-speaking with at least one English-speaking parent
* 5. vitamin D deficiency (<20 ng/mL)
* 6. compliant with attending at least 2/4 of their last asthma-related scheduled clinic visits

Exclusion Criteria:

* 1. If female, pregnant, planning to become pregnant, and/or sexually active and not using reliable contraception
* 2. Unable to provide informed consent (mental retardation, etc)
* 3. Current substance dependence (within the past 2 months)
* 4. Known metabolic bone disease, including rickets
* 5. Known malabsorption disease: Crohn's, ulcerative colitis, celiac sprue
* 6. BMI>40
* 7. Has begun new treatment with vitamin D (>600 IU/day) within the past month
* 8. Treatment with prednisone or other oral or IV steroid within the past 4 weeks
* 9. Taking mineral oil or thiazide diuretics on a daily basis
* 10. Acute or chronic liver, renal, endocrine, neurologic, infectious, autoimmune, cardiac, pulmonary, gastrointestinal, hematologic, metabolic disorder or any other disorder, per study physician judgment.
* 11. Severe treatment noncompliance documented in medical record or by managing provider report.

Our definition of a highly effective method of birth control is consistent with ICH Guidance for Industry M3 Nonclinical Safety Studies for the Conduct of Human Clinical Trials for Pharmaceuticals (April 1997) when used consistently and correctly, such as implants, injectables, oral contraceptives, some intrauterine devices (IUDs), sexual abstinence, or a vasectomized partner. Subjects will also be reminded to use condoms to prevent sexually transmitted diseases and as a second method toward birth control.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
vitamin D levels | change in serum vitamin D level from baseline to 12 weeks
  Primary:
  1. 25-OH vitamin D (D2, D3): 1.0 ml sample sent to Esoterix Laboratory Services (Austin, TX) through NCH and run via high pressure liquid chromatography (HPLC), Tandem Mass Spectrometry analysis. Samples processed individually, not batched, for intervention study purposes.

SECONDARY OUTCOMES:
Side Effects Form for Children and Adolescents (SEFCA) | Baseline, end of week 12
  structured interviewer-administered questionnaire inquiring about body systems health and concerns
Block Kids 2004 Food Frequency Questionnaire | baseline, and end of week 12
  a questionnaire inquiring how often children eat particular items from different food groups
immune status | baseline, and end of week 12
  key pro-inflammatory and anti-inflammatory cytokines as well as T-cell ratios will be compared before and after vitamin D supplementation

OTHER OUTCOMES:
asthma severity | baseline, and end of week 12
  via pulmonary function tests
quality of life | Baseline, and end of week 12
  pediatric quality of life questionnaire, including questions about asthma
omega fatty acid profile | Baseline, and end of week 12
  red blood cells will be analyzed for omega fatty acid percentages and ratios of omega 3 fatty acids will be compared to omega 6 fatty acids.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Gracious, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States